CLINICAL TRIAL: NCT01034891
Title: Women At Risk: The High Risk Breast Cancer Program
Acronym: WAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: New York Presbyterian Hospital (Other)
Collaborators: Women At Risk (Ambiguous)
Responsible Party: Amy Whiffen, Women At Risk
Other Study IDs: AAAA4649
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-10

CONDITIONS: Breast Cancer
Keywords: BRCA mutation; benign breast disease; family history of breast cancer; strong family history of breast cancer; atypical ductal hyperplasia; atypical lobular hyperplasia; high risk for breast cancer
MeSH Terms: conditions — Breast Neoplasms; Cystic Fibrosis; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to increase understanding of women who are at high risk for developing breast cancer. Data from this group will be collected and entered into a registry. This registry serves as a clinical database to support research in prevention, early detection and treatment of breast cancer.

DETAILED DESCRIPTION:
This is a longitudinal cohort study that collects data of eligible women at risk for developing breast cancer. Patient information will be entered into a secured computerized database that is used for research on the prevention, early detection and treatment of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* one or more first-degree relatives (mother, daughter, or sister) with pre-menopausal breast cancer
* two or more first-degree relatives with post-menopausal breast cancer
* tested positive for a BRCA1 or BRCA2 mutation
* a history of biopsy-proven atypical ductal hyperplasia or atypical lobular hyperplasia
* a history of biopsy-proven lobular neoplasia (lobular carcinoma in situ)

Exclusion Criteria:

* DCIS (ductal carcinoma in situ)
* previous diagnosis of breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of the breast center at New York Presbyterian Hosptial/ Columbia University Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 1991-01

CONTACTS AND LOCATIONS:
Overall Officials: Kathie-Ann Joseph, MD, MPH, Principal Investigator — Columbia University/New York Presbyterian Hospital
Locations (2):
- United States (2):
  - Women At Risk, Columbia University Medical Center, New York, New York
  - Women At Risk, Weill Cornell, New York, New York

REFERENCES:
- [Result] Chun J, Pocock B, Joseph KA, El-Tamer M, Klein L, Schnabel F. Breast cancer risk factors in younger and older women. Ann Surg Oncol. 2009 Jan;16(1):96-9. doi: 10.1245/s10434-008-0176-8. Epub 2008 Nov 1. PMID 18979140
- See also: Women At Risk Website — http://nyp.org/services/war/index.html